CLINICAL TRIAL: NCT06507410
Title: Additive Effects of Clonidine Used in Propofol Sedation in Colonoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rabab Mohamed Mohamed Mohamed, Assistant Professor of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR725/6/24
Record Dates: First submitted 2024-07-11; First posted 2024-07-18 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Clonidine; Propofol; Sedation; Colonoscopy
MeSH Terms: interventions — Propofol; Clonidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol group (Active Comparator): Patients will receive induction of sedation as follow:
  Continuous propofol infusion will be given with syringe pump for maintenance, with the initial rate set at 25-75 mic/kg/min IV during the first 10-15 min. To avoid administering sedatives at rates greater than clinically necessary, infusion rates will be gradually titrated to 25-50 mic/kg/min and regulated with the clinical response, with an onset of peak drug action expected to occur within 2 min.
  Interventions: Drug: Propofol
- Propofol combined with clonidine group (Experimental): Patients will receive 2 μg/kg of clonidine for injection intravenously 30 min before induction of sedation, administered over 10 min.
  Interventions: Drug: Propofol combined with clonidine

INTERVENTIONS:
Drug: Propofol — Continuous propofol infusion will be given with syringe pump for maintenance, with the initial rate set at 25-75 mic/kg/min IV during the first 10-15 min. To avoid administering sedatives at rates greater than clinically necessary, infusion rates will be gradually titrated to 25-50 mic/kg/min and regulated with the clinical response, with an onset of peak drug action expected to occur within 2 min.
  Arms: Propofol group
Drug: Propofol combined with clonidine — Patients will receive 2 μg/kg of clonidine for injection intravenously 30 min before induction of sedation, administered over 10 min.
  Arms: Propofol combined with clonidine group

SUMMARY:
The objective of this study was to compare safety, satisfaction, and efficiency outcomes of propofol versus propofol with clonidine in patients undergoing colonoscopy.

DETAILED DESCRIPTION:
Colonoscopy is one of the most common procedures in the world, Colonoscopy is a procedure often performed for prevention, diagnosis, and treatment of a variety of symptoms and diseases of the lower digestive tract, and sedation or anesthesia should be considered as an important tool to increase its effectiveness.

Sedation and analgesia are considered key components, as they reduce anxiety and discomfort and therefore improve the procedure tolerability and patient satisfaction, minimize risk of complications and provide better conditions for the examination.

Propofol may be used alone or in combination with opioids and/or benzodiazepines.

The use of propofol alone requires higher doses, which may lead to increased incidence of side effects. However, the risks and benefits of adding analgesic and sedative to propofol are controversial, and the selection of drugs is a crucial factor in determining the outcomes.

Clonidine apparently produces its sedative and anaesthetic-sparing effects by stimulation of centrally located alpha2 adrenoceptors. Analgesia seems to be mediated mainly by activation of alpha2 adrenoceptors in the dorsal horn of the spinal cord.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Patients undergoing colonoscopy.

Exclusion Criteria:

* Patients had recent history of colonoscopy.
* Previous colonic resection.
* Severe heart failure (ejection fraction < 30%).
* Known history of hypersensitivity to propofol or clonidine and any need for anesthetic drug administration other than the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 24 hours postoperatively
  Patient's satisfaction level will be assessed with a Likert five-item scoring system (1 = Not at all satisfied, 2 = slightly satisfied, 3 = somewhat satisfied, 4 = very satisfied, and 5 = extremely satisfied).

SECONDARY OUTCOMES:
Heart rate | Till the end of surgery
  Heart rate will be recorded at 30 minutes before induction, at induction, and at the end of surgery.
Mean arterial blood pressure | Till the end of surgery
  Mean arterial blood pressure will be recorded at 30 minutes before induction, at induction, and at the end of surgery.
Side effects | 24 hours postoperatively
  Side effects such as nausea and vomiting, psychological reactions will be noted.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.